CLINICAL TRIAL: NCT03188276
Title: The Relationship Between Direct Acting Antiviral Treatment Effect and Myeloid-Derived Suppressor Cells and NK Cells Activity in Chronic Hepatitis C
Brief Title: The Relationship Between MDSCs and NK Cells Activity of CHC Patient Treated by DAAs
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chao-Shuang Lin, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Effect of DAAs on MDSCs and NK
Record Dates: First submitted 2017-06-11; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; direct-acting antiviral agents; Myeloid-Derived Suppressor Cells; NK cells
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ledipasvir, sofosbuvir drug combination; daclatasvir

STUDY DESIGN:
Intervention Model Description: There are 32 treatment-naive CHC patients who treated by Ledipasvir-Sofosbuvir or Daclatasvir-Sofosbuvir.
Masking Description: Thr care provider, participant, investigator and outcomes assessor all konw the process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHC patients (Active Comparator): 32 treatment-naive CHC patients treated by Ledipasvir-Sofosbuvir or Daclatasvir-Sofosbuvir.
  Interventions: Drug: Ledipasvir-Sofosbuvir; Drug: Daclatasvir-Sofosbuvir
- Healthy controls (No Intervention): 20 Healthy controls without any treatment

INTERVENTIONS:
Drug: Ledipasvir-Sofosbuvir — 15 CHC patients were treated with Sofosbuvir (400mg, qd)/Ledipasvir (90mg, qd) for 12 weeks
  Other Names: Harvoni
  Arms: CHC patients
Drug: Daclatasvir-Sofosbuvir — 17 CHC patients were treated with Sofosbuvir (400mg, qd)/Daclatasvir (60mg,qd) for 12 weeks.
  Other Names: Daklinza
  Arms: CHC patients

SUMMARY:
Hepatitis C virus (HCV) infection is easy to chronic and can progress to cirrhosis and liver cancer. Direct-acting antiviral treatment can significantly improve the prognosis of the disease and the efficacy is seemingly not affected by a variety of viral factors. In addition, direct-acting antiviral agents therapy may affect the transformation of the immune cells and ameliorate the host immune status consequently. This study mainly investigated the relationship between Direct Acting Antiviral Treatment effect and the functional activity of myeloid-derived suppressor cells (MDSCs) and natural killer cells (NK cells) in Chronic Hepatitis C.

DETAILED DESCRIPTION:
32 treatment-naive CHC patients and 20 healthy controls were recruited. Patients were examined before DAAs therapy (0w) and at weeks 4 (4w) and weeks 12 (12w) and weeks24 (24w) of the therapy. The percent age of myeloid-derived suppressor cells and NK cells of the peripheral blood were analyzed by flow cytometry. The investigators discuss the relationship between direct acting antiviral treatment effect and myeloid-derived suppressor cells and NK cells activity in chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Positive serum Anti-HCV antibody or serum HCV-RNA, CHC patients without any treatment

Exclusion Criteria:

* Patient has a history of clinical signs/symptoms of hepatic decompensation (Child-Pugh Grade B or C) or ascites, esophageal variceal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis.
* Patient has a history of hepatocellular carcinoma (HCC) or suspected symptoms of HCC, such as suspicious foci on imaging studies and/or serum alpha-fetoprotein (AFP)>50ng/mL.
* Patient has received IFN or other immunomodulatory treatment within 52 weeks before Screening.

Patient has a medical condition that requires frequent use of systemic acyclovir or famciclovir.

* Patient has a medical condition that requires frequent use of systemic corticosteroids, however topical and inhaled corticosteroids are allowed.

Patient has used hepatotoxic drugs within one month. Patient has overtaken alcohol (>40g/day) or abused illicit drugs in recent one year.

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test.
* Patients who co-infected with HAV, HBV, HDV, HEV,HIV(human immunodeficiency virus ) Patient has one or more additional known primary or secondary causes of liver disease, other than hepatitis C (e.g., alcoholism, autoimmune hepatitis).

History of malignancy of any organ system.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Changes of the frequency of CD14+CD11b+CD33+HLA-DR-/low MDSCs | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of CD14+CD11b+CD33+HLA-DR-/low MDSCs of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)

SECONDARY OUTCOMES:
Changes of the frequency of CD14+HLA-DR-/low M-MDSCs | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of CD14+HLA-DR-/low M-MDSCs of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)
Changes of the frequency of CD3+CD4+ T cells | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of CD3+CD4+ T cells of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)
Changes of the frequency of CD3+CD8+ T cells | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of CD3+CD8+ T cells of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)
Changes of the frequency of CD3CD56+ NK cells | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of CD3CD56+ NK cells of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)
Changes of the frequency of NKG2A in CD3CD56+ NK cells | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of NKG2A in CD3CD56+ NK cells of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)
Changes of the frequency of NKp30 in CD3CD56+ NK cells | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of NKp30 in CD3CD56+ NK cells of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)
Changes of the frequency of NKp46 in CD3CD56+ NK cells | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks ( 24 weeks after DAAs treatment)
  Measurement of the frequency of NKp46 in CD3CD56+ NK cells of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment), 12 weeks (12 weeks after DAAs treatment) and 24 weeks (24 weeks after DAAs treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-liang Gao, PhD, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not available to other researchers